CLINICAL TRIAL: NCT01354665
Title: The Short-term Effect of Immunomodulatory Treatment With Interferon Beta-1b (Betaferon) on Fatigue and Depression in First-time Treated Patients With Relapsing-remitting Multiple Sclerosis.
Brief Title: Depression and Fatigue in MS Patients Treated With Betaferon.
Acronym: FADO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15307; BF1012PL (Other: NIS Trial Alias)
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Interferon beta-1b; Fatigue; Depression
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Depression | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Biological: Interferon beta-1b (Betaferon, BAY86-5046)

INTERVENTIONS:
Biological: Interferon beta-1b (Betaferon, BAY86-5046) — Patients treated with regular dose of Betaferon injections (250 micrograms subcutaneously every other day) under routine practice setting.

SUMMARY:
This study aims to evaluate the occurence and severity of fatigue and depression in multiple sclerosis patients and the impact of Betaferon treatment on symptoms alterations.

The study is conducted in routine practice setting hence no interference with standard care takes place.

Pharmacologic treatments of MS-fatigue and depression will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting multiple sclerosis
* Age 18+
* Patients initiating Betaferon treatment

Exclusion Criteria:

* Patients previously treated with any immunomodulatory drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with relapsing form of multiple sclerosis treated with Betaferon under routine practice setting.
Sampling Method: Probability Sample
Enrollment: 567 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Changes of fatigue score over time | short-term, mid-term and long-term changes will be assessed: 3 months vs. baseline, 6 months vs. baseline and 12 months vs. baseline

SECONDARY OUTCOMES:
Changes of depression score over time | short-term, mid-term and long-term changes will be assessed: 3 months vs. baseline, 6 months vs. baseline and 12 months vs. baseline
Treatment adherence | 12 months
Clinical course of the disease | 12 months
Overall treatment tolerability as measured by rate of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland